CLINICAL TRIAL: NCT00863733
Title: Phase I Trial of 5,6 Dimethylxanthenone - 4 - Acetic Acid (DMXAA) in Solid Tumors
Brief Title: Study of DMXAA (Now Known as ASA404) in Solid Tumors
Acronym: DMXAA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: Cancer Society Auckland (Other)
Responsible Party: Dr Paul Thompson, Auckland Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHI/050
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Solid Tumors
MeSH Terms: interventions — vadimezan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: DMXAA — Administered as a 20 minute IV infusion, once every three weeks at doses ranging from 6 mg/m2 to 4900 mg/m2
  Other Names: 5,6 Dimethylxanthenone-4-Acetic Acid; ASA404; AS1404; NSC-640488

SUMMARY:
This is a phase I study aimed at identifying safe doses of DMXAA in patients with solid tumors.

DETAILED DESCRIPTION:
This is a dose escalation study conducted at a single center in New Zealand. Patients received dimethylxanthenone acetic acid (DMXAA) IV over 20 minutes once every three weeks, up to a maximum of 12 courses.

Cohorts of 3 patients received escalated doses of DMXAA until the maximum tolerated dose (MTD) was determined. The MTD is defined as the dose preceding that at which 2 of 3 patients experience dose limiting toxicity.

Patients had solid tumors for which there was no standard therapy or were refractory to conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed solid tumor that is not amenable to any standard therapy or is refractory to conventional therapy
2. Performance status WHO 0-2
3. Life expectancy greater than 3 months
4. Hemoglobin at least 90 g/L; WBC at least 3,000/mm3; Platelet count at least 100,000/mm3
5. Bilirubin within normal limits; ALT less than 2 times upper limit of normal (ULN); Alkaline phosphatase less than 2 times ULN
6. Creatinine less than 130 umol/L
7. INR and APTT within normal limits
8. Fertile patients must use effective contraception
9. At least 4 weeks since prior anticancer therapy and recovered from toxic effects

Exclusion Criteria:

1. Concurrent malignancy except cone biopsied carcinoma in situ of the cervix and adequately treated basal or squamous cell carcinoma of the skin
2. Other serious medical condition
3. Uncontrolled infection or serious infection within the past 28 days
4. Pregnant or lactating
5. Treatment with glucocorticosteroids within previous two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 1996-05; Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Toxicity of DMXAA
Maximum tolerated dose of DMXAA
Pharmacokinetics of DMXAA
Effect of DMXAA on coagulation parameters, TNF and other cytokine production, nitric oxide, and serotonin production

SECONDARY OUTCOMES:
Efficacy of DMXAA
Effect of DMXAA on tumor vasculature

CONTACTS AND LOCATIONS:
Overall Officials: Dr Paul Thompson, Principal Investigator — Auckland Hospital

REFERENCES:
- [Result] Jameson MB, Thompson PI, Baguley BC, Evans BD, Harvey VJ, Porter DJ, McCrystal MR, Small M, Bellenger K, Gumbrell L, Halbert GW, Kestell P; Phase I/II Trials Committee of Cancer Research UK. Clinical aspects of a phase I trial of 5,6-dimethylxanthenone-4-acetic acid (DMXAA), a novel antivascular agent. Br J Cancer. 2003 Jun 16;88(12):1844-50. doi: 10.1038/sj.bjc.6600992. PMID 12799625
- [Derived] Jameson MB, Sharp DM, Sissingh JI, Hogg CR, Thompson PI, McKeage MJ, Jeffery M, Waller S, Acton G, Green C, Baguley BC. Transient retinal effects of 5,6-dimethylxanthenone-4-acetic acid (DMXAA, ASA404), an antitumor vascular-disrupting agent in phase I clinical trials. Invest Ophthalmol Vis Sci. 2009 Jun;50(6):2553-9. doi: 10.1167/iovs.08-2068. Epub 2009 Apr 22. PMID 19387077